CLINICAL TRIAL: NCT02044692
Title: The Long-term Safety of Hunterase (Idursulfase-beta) in Hunter Syndrome(Mucopolysaccharidosis II) Patients
Brief Title: The Long-term Safety Study of Idursulfase-beta in Hunter Syndrome(Mucopolysaccharidosis II) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Other Study IDs: GC1111_OS
Record Dates: First submitted 2014-01-19; First posted 2014-01-24 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Hunter Syndrome
Keywords: Hunter syndrome; Mucopolysaccharidosis II; Hunterase
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the long term safety and efficacy of once weekly dosing of idurasulfase-beta 0.5mg/kg administered in Hunter Syndrome(Mucopolysaccharidosis II) Patients

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a diagnosis of Hunter syndrome(Mucopolysaccharidosis II).
* Patients who are administered idurasulfase-beta or willing to be administered idurasulfase-beta.
* Patient's parent(s), or patient's legal guardian must have given voluntary written consent to participate in the study.

Exclusion Criteria:

* Patients who have participated in any other blind clinical trials.
* Patient who cannot be tracked about safety.
* Patients who are judged disqualified to participate clinical trials by investigator for other causes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hunter Syndrome(Mucopolysaccharidosis II) Patients
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event and adverse drug reaction. | Once a week up to 5years

SECONDARY OUTCOMES:
Change of vital sign, physical and clinical examination, anti-idurasulfase-beta antibody status. | Base line and every three months up to 5years.(exception: clinical examination-> baseline and every six months up to 5years)

OTHER OUTCOMES:
Percent change of urine GAG. | Baseline and every three months up to 5years.
Percent change of 6 minute walking test. | Baseline and every 6 months up to 5years.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Kyu Jin, Principal Investigator — Samsung medical center, Seoul, Republic of Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea